CLINICAL TRIAL: NCT05946928
Title: CLINICAL EVALUATION AND IMPACT ON EMERGENCE AGITATION OF AN ORAL SOLUTION OF MIDAZOLAM CONTAINING g-CICLODEXSTRIN IN PAEDIATRIC MAGNETIC RESONANCE IMAGING: A RETROSPECTIVE COHORT STUDY
Brief Title: EMERGENCE AGITATION After Premedication IN PAEDIATRIC MAGNETIC RESONANCE IMAGING: A RETROSPECTIVE COHORT STUDY
Acronym: premidazolam
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Garra Rossella, Medical doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 0032517/22
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Autism Spectrum Disorder; Premedication; Brain Neoplasms; Brain Pathology; Growth Retardation
MeSH Terms: conditions — Autism Spectrum Disorder; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ozased group: 50 patients premedicated with OZALIN® / OZASED®
- Control group: 50 patients who did not receive any premedication

SUMMARY:
The aim of this study was to assess the anxiolytic and sedative effect of OZALIN® / OZASED® (ADV6209) 0,25mg/Kg in children undergoing magnetic resonance imaging (MRI) under inhalational anesthesia. Our hypothesis is that compared to children who do not receive any premedication, palatability of OZALIN® / OZASED® by allowing an easier acceptance of the drug, improves the quality of anesthesia induction and postoperative behavioral outcome improving sedation and reducing the need for inhalation anesthetic which has been recognized as the main cause of post-procedural behavioral changes, including emergence agitation.

DETAILED DESCRIPTION:
Magnetic resonance imaging is considered the primary investigative tool for evaluating a wide range of paediatric medical conditions. Sedatives are often needed in this population to ensure immobilization during the acquisition of the images.

Midazolam has always been the most used anxiolytic-sedative drug in the pediatric population. Over time, the intravenous formulation of midazolam has been used also for oral, nasal or rectal administration but those alternative routes of administration represent an off-label use. Recently, in Europe was licensed ADV6209, a midazolam solution for oral use containing gamma-cyclodextrin (OZALIN® / OZASED®).

The aim of this study was to assess its anxiolytic and sedative effect at a dosage of 0,25mg/Kg in children undergoing magnetic resonance imaging (MRI) under inhalational anesthesia. Our hypothesis is that compared to children who do not receive any premedication, palatability of OZALIN® / OZASED® by allowing an easier acceptance of the drug, improves the quality of anesthesia induction and postoperative behavioral outcome improving sedation and reducing the need for inhalation anesthetic which has been recognized as the main cause of post-procedural behavioral changes, including emergence agitation.

ELIGIBILITY:
Inclusion Criteria:

- We included in the study 100 children (either gender), aged 1-10 years, American Society of Anaesthesiologists (ASA) physical status 1 and 3 who, between March and December 2022, received inhalation anesthesia for brain and spinal cord MRI for diagnostic investigations or postoperative and oncological follow-up

Exclusion Criteria:

* 1) a history of hypersensitivity to midazolam; 2) chronic therapy with benzodiazepines; 3) acute respiratory tract infections; 4) psychiatric and behavioural disorders; 5) ASA physical status >3.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: the IRCCS Agostino Gemelli Foundation of Catholic University of Rome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
evaluation of patients' reactive behavior to facemask positioning for inhalational anesthesia induction. | 30 minutes within premedication administration
  evaluation of patients' reactive behavior to facemask positioning for inhalational anesthesia induction evaluated on a four-point scale (Mask Acceptance Scale, MAS) indicating that child is cooperative and accept the mask readily (MAS=1), he is slight fearful and accepts the mask with mild resistance (MAS=2), with moderate struggle (MAS=3) or he resists strongly and must be restrained (MAS=4)

SECONDARY OUTCOMES:
the percentage of sevoflurane at which the child's eyes closed upon induction of general anesthesia | procedure (at induction of general anesthesia)
  the percentage of sevoflurane at which the child's eyes closed upon induction of general anesthesia;
time to eye closure at induction of anesthesia; | procedure (at induction of general anesthesia)
  time to eye closure at induction of anesthesia
patient degree of acceptance of the administered premedication | 30 minutes before induction of general anesthesia
  degree of acceptance of the administered premedication
evaluation of OZALIN® / OZASED® anxiolytic efficacy | 30 minutes after premedication administration
  OZALIN® / OZASED® anxiolytic efficacy was evaluated 30 minutes after premedication administration with the Ramsay sedation scale
child's behavior on separation from the parent | baseline (before induction of general anesthesia)
  Child's behavior at the moment of separation from the parent just before induction of anesthesia was evaluated with a four-point Parental Separation Anxiety scale (PSAS)
occurrence of delirium at the emergence from anesthesia | at emergence of anesthesia procedure
  The occurrence of emergence delirium at the end of the procedure was measured using the five items of the Pediatric Anesthesia Emergence Delirium scale (PAED)
evaluation of behavioural changes seven days after the procedure, between the two groups. | 7 days after the magnetic resonance Imaging
  Maladaptive behavioural responses and developmental regression seven days after the procedure were evaluated by parents of children with the Post Hospitalization Behaviour Questionnaire for Ambulatory Surgery (PHBS-AS).

CONTACTS AND LOCATIONS:
Overall Officials: Rossella Garra, Principal Investigator — Fondazione Policlinico A. gemelli IRCCS
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Non completely planned yet
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Non completely planned yet
Access Criteria: Not completely planned yet